CLINICAL TRIAL: NCT04086420
Title: A Mindfulness-Based Physical Activity Intervention: A Randomized Pilot Study
Brief Title: Mindfulness-Based Physical Activity Intervention
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H18-046 SALM
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Mindfulness; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Mindfulness; Heart Rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Delivered through an audio-recording consisting of a single meditation exercise that lasted for 30 minutes
  Interventions: Behavioral: Mindfulness
- Heart-Rate (Active Comparator): Given a heart rate monitor and instructed to use it to determine the intensity of their exercise
  Interventions: Behavioral: Heart-Rate

INTERVENTIONS:
Behavioral: Mindfulness — Received instructions to exercise at moderate intensity while listening to an audio-recorded mindfulness-based physical activity intervention
  Arms: Mindfulness
Behavioral: Heart-Rate — Given a heart rate monitor, told to exercise within the moderate intensity range (64-76% of estimated maximum heart rate)
  Arms: Heart-Rate

SUMMARY:
The aims of this parallel two-arm pilot randomized controlled trial is to assess the feasibility and acceptability of an audio-recorded mindfulness-based intervention and to assess whether the intervention results in a clinically meaningful difference in physical activity compared to the control condition

ELIGIBILITY:
Inclusion Criteria:

* Reported less than 60-minutes of weekly moderate-to-vigorous physical activity (MVPA, moderate physical activity minutes + vigorous physical activity minutes*2)
* Safe to exercise at moderate intensity without a doctor's approval according to American College of Sports Medicine Criteria
* Had a smart phone to access the audio-recorded mindfulness-based physical activity intervention

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity Minutes | 1-Week Follow-Up

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Methodist University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sala M, Geary B, Baldwin AS. A Mindfulness-Based Physical Activity Intervention: A Randomized Pilot Study. Psychosom Med. 2021 Jul-Aug 01;83(6):615-623. doi: 10.1097/PSY.0000000000000885. PMID 33165218